CLINICAL TRIAL: NCT03186911
Title: The Impact of E-liquid Nicotine Content on Reinforcement in Current Smokers
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Study team decided not to move forward with study
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: U54 DA031659-06 Pilot; 1U54DA031659-01 (NIH)
Record Dates: First submitted 2017-06-08; First posted 2017-06-14 (Actual); Last update posted 2019-08-05 (Actual); Status verified 2018-10

CONDITIONS: Tobacco Use
MeSH Terms: conditions — Tobacco Use

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- E-liquid Group (Other): Participants will sample two different e-liquids.
  Interventions: Behavioral: E-liquid sampling and preference assessment

INTERVENTIONS:
Behavioral: E-liquid sampling and preference assessment — Participants will sample two different e-liquids that vary in nicotine content, complete questionnaires about each one, and then choose between the two e-liquids in a preference assessment task.

SUMMARY:
Participants will complete a phone screen and then one laboratory session. After completing in-person screening assessments, eligible participants will complete additional questionnaires. Participants will then choose an e-liquid flavor to use for the rest of the session. Participants will then sample two e-liquids that vary in nicotine content from little or no nicotine to a moderate level of nicotine, and questionnaires evaluating the subjective effects of each one. Participants will then complete a preference assessment where they choose between the two e-liquids. Participants will be blind to the nicotine contents.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years old
* Daily cigarette smoking
* Have tried vaping devices on a minimum of one lifetime occasion

Exclusion Criteria:

* Unwilling to use a vaping device during the session
* Break alcohol level > 0.01 (g/dL)
* Pregnant, trying to become pregnant, or breastfeeding
* Systolic BP greater than or equal to 160 mm/Hg or below 90 mm/Hg
* Diastolic BP greater than or equal to 100 mm/Hg or below 50 mm/Hg
* Heart rate greater than or equal to 105 bpm or lower than 45 bpm
* A current upper respiratory infection, recent cardiac event (in the last year), Buerger disease, irregular heartbeat or arrhythmia within the last year, previous allergic or adverse reaction to nicotine

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-07 (Estimated); Primary Completion 2019-09 (Estimated); Study Completion 2019-09 (Estimated)

PRIMARY OUTCOMES:
Product Evaluation Questionnaire | One Day
  Ratings of the two e-liquids on a self-report questionnaire

SECONDARY OUTCOMES:
Preference Assessment | One Day
  Choices of each of the two e-liquids on a preference assessment
Perceived Health Risk Questionnaire | One Day
  Personal Health Risk Ratings about each of the two e-liquids
Vaping Purchase Task | One Day
  Hypothetical estimates of consumption of each of the e-liquids across a variety of prices

CONTACTS AND LOCATIONS:
Overall Officials: Eric C Donny, PhD, Principal Investigator — Wake Forest University Health Sciences

IPD SHARING:
Plan to Share IPD: No